CLINICAL TRIAL: NCT01493661
Title: Chronic Sleep Restriction: Neurobehavioral and Physiological Responses
Brief Title: Chronic Sleep Restriction
Acronym: CSR
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marco Tulio de Mello, Ph.D, Federal University of São Paulo
Other Study IDs: CEPE2011SSQueiroz
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Other Conditions That May Be A Focus of Clinical Attention
Keywords: Sleep; Polysomnography; Reaction Time; Sleep Deprivation; Psychophysiology; Chronic sleep restriction; healthy; without sleep complaints
MeSH Terms: conditions — Sleep Deprivation | interventions — Sleep

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Men with Total Sleep Time ≤ 6h that will undergo 25 percent of chronic sleep restriction of their TST
  Interventions: Other: Chronic Sleep Restriction
- Group 2: Men with Total Sleep Time (range 7-8h)that will undergo 25 percent of chronic sleep restriction of their TST
  Interventions: Other: Chronic Sleep Restriction
- Group 3: Men with Total Sleep Time ≥ 9h that will undergo 25 percent of chronic sleep restriction of their TST
  Interventions: Other: Chronic Sleep Restriction

INTERVENTIONS:
Other: Chronic Sleep Restriction — All volunteers will undergo 25% of sleep restriction of their total sleep time at the beginning sleep for five consecutive days. The nights will be monitored by polysomnography.
  Other Names: Chronic; Sleep; Restriction

SUMMARY:
Sleep is a physiological state considered essential for health and human survival. The prevalence of chronic sleep restriction has increased in modern society, as well as the effects of the same health concerns about various aspects, including the physiological and neurobehavioral. The objective of this study is to identify the neurobehavioral and physiological responses of healthy men with different needs of total sleep time (TST) submitted to chronic sleep restriction. Participants in this study will be 30 male volunteers, aged between 20 and 35 years, divided into three groups: Group 1 (n = 10) with TST ≤ 6 hours (h), Group 2 (n = 10) with TST ≥ 9h and Group 3 (n = 10): TST with between 7 and 8h. The TST will be established by the constant and continuous use of actigraphy for 10 days prior to the onset of the experimental protocol. All volunteers will undergo medical and polysomnography (PSG) examination to detect the presence or not of changes in sleep as well as other health problem that prevents their participation in the study. The experimental protocol consists of a basal night of sleep, five consecutive nights of chronic sleep restriction to 25% of TST in the beginning night and a night of recovery, which will be allowed to sleep the sleep pattern. Each night will have PSG monitoring and when wake up in each day, the volunteer will undergo tests to assess the physiological and neurobehavioral variables. The significance level will be 5% (p ≤ 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≤ 25 kg/m2
* Physically active individuals
* 8 years of school education.

Exclusion Criteria:

* High level of anxiety - State-Trait Anxiety Inventory (STAI-T) ≥ 35
* High level of anxiety - Beck Depression Inventory ≥ 19
* PSQI - Pittsburgh Sleep Quality Index ≥ 11
* ESS - Epworth Sleepiness Scale ≥ 15
* Irregular rhythm of sleep identified by actigraphy
* Sleep disturbance by polysomnography
* Shift worker or nocturnal worker;
* Obesity;
* Smoker;
* Alcohol Intake of more than 3 drinks per day;
* Taking sleep medications or illicit drugs.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample, residents of Sao Paulo city
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco T De Mello, Ph.D, Principal Investigator — Federal University of São Paulo; Juliana MS Prado, Ph.D, Study Chair — Federal University of São Paulo; Patricia Rzezak, Ph.D, Study Chair — Federal University of São Paulo; Sergio Tufik, Ph.D, Study Chair — Federal University of São Paulo; Sandra S De Queiroz, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Fundação de Amparo à Pesquisa do Estado de São Paulo — http://www.fapesp.br/